CLINICAL TRIAL: NCT04355923
Title: Impact of Confinement on the Treatment of Spondyloarthritis.
Brief Title: Confinement and Spondyloarthritis Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20rhumatocovid01
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the impact of confinement on treatment use in spondyloarthritis. Study hypothesis that with the confinement, subjects will stop their treatment. The main objective is to study the impact of confinement on treatment. And secondly to look for for specific psychological profile linked to the interruption of the treatment. the study population consists of patients with spondyloarthritis and belonging to a patient association (ACS). All patients over 18 are included. A mailing questionnaire will be send to all patients. data on diseases activity and treatment will be collected

ELIGIBILITY:
Inclusion Criteria:

* spondyloarthritis,
* age over 18 ans
* treatment by NSAID or biological treatment to be part of the patient association "ACS" (action contre les spondylarthropathies).

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with spondyloarthritis and member of ACS patient association group
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
treatment use | 1 month
  treatment continuation

SECONDARY OUTCOMES:
activity of disease | 1 week
  number of crisis
psychological aspects | 1 month
  Ten Item Personality Inventory rated on a scale from 1, disagree strongly, to 7, agree strongly)
psychological aspects | 1 month
  quality of life questionnaire (EQ-5D) evaluating mobility, self care, usual activity, pain and anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established